CLINICAL TRIAL: NCT01792271
Title: Novel Therapies for Muco-Obstructive Lung Diseases: Sustained Effects of Hypertonic Saline on Mucociliary Clearance and Clinical Tolerability in Subjects With Chronic Bronchitis
Brief Title: Sustained Effects of Hypertonic Saline on Mucociliary Clearance in Subjects With Chronic Bronchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 12-2602; 1P01HL108808-01A1 (NIH)
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Chronic Obstructive Pulmonary Disease; COPD; Chronic Bronchitis
Keywords: COPD; Chronic Bronchitis; Hypertonic Saline
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic | interventions — Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AB: 7% HS home tx, then 0.12% NaCl (Placebo Comparator): Inhaled Inhaled 7% HS (hypertonic saline) home treatment' , then 0.12% sodium chloride solution home treatment.
  The intervention consists of the subject receiving both concentrations of inhaled sodium chloride solution, each during a different home treatment periods. Subjects randomized to order AB will receive inhaled 7% NaCl (sodium chloride solution) mist during the first home treatment period, then 0.12% NaCL during the second home treatment period.
  Interventions: Other: Inhaled 7% HS (NaCl) home treatment
- BA: 0.12% NaCl home tx, then 7% HS (Placebo Comparator): Subjects randomized to order BA will receive inhaled 0.12% NaCl mist during the first home treatment period, then Inhaled 7% HS home treatment during the second home treatment period.
  Interventions: Other: Inhaled 7% HS (NaCl) home treatment

INTERVENTIONS:
Other: Inhaled 7% HS (NaCl) home treatment — Administering inhaled 7% NaCl for two weeks of home treatment vs. a placebo of 0.12% NaCL during a separate home treatment period, and assessing the effects of each primarily by MCC study.

SUMMARY:
The purpose of this research study is to examine the effects of two weeks of daily dosing of inhaled salt water mist (hypertonic saline - HS) on actual measurements of mucociliary and cough clearance in patients with the chronic bronchitis type of Chronic Obstructive Pulmonary Disease (COPD.

Defective mucociliary clearance (MCC) is central to the development and/or worsening of several kinds of lung diseases, including COPD/chronic bronchitis (CB), cystic fibrosis (CF), and bronchiectasis. In each case, defective MCC leads to the development of lung infections and damage to the airways from ongoing inflammation caused by a person's inability to clear mucus from the lungs.

The investigators' previous studies have shown that the administration of inhaled HS (hypertonic saline) not only acutely accelerates MCC in CF, but also that repetitive use "resets" the baseline rate of MCC within 2 weeks. It is likely that the sustained effect of HS on MCC was responsible for the ~60% reduction in the frequency of pulmonary disease exacerbations, reduced antibiotic use and improved lung function in a long-term study of HS in CF volunteers. As a result, HS has now become a standard therapy for CF lung disease and its success raises optimism that similar benefits might occur in patients with CB.

In this study the investigators will use mildly radioactive particles, technetium bound to sulfur colloid, to measure and compare the sustained effects on mucus clearance of two weeks of daily dosing of 7% hypertonic saline versus a low salt control treatment for subjects with CB. We will also be collecting sputum and breath condensation to analyze for protein and inflammatory changes that might occur with exacerbations.

Our long term goals are to improve our understanding of MCC in health and disease and to develop better therapies that support and/or restore MCC in patients with these diseases to reduce lung infections.

ELIGIBILITY:
Inclusion Criteria:

Volunteers who meet all of the following criteria will be eligible for study participation:

1. Age 40-80 years, inclusive
2. Non-pregnant subjects must be either not sexually active, post-menopausal, surgically sterilized, or agree to use an appropriate "double barrier" method (such as diaphragm and condom), or must currently be using a prescribed transdermal, injection, implant, or oral contraceptive during study participation.
3. Forced expiratory volume in 1 second (FEV1) of 35-80% of predicted, inclusive, and FEV1/forced vital capacity (FVC) < 70%
4. Produces mucus at least 2 days per week, on average
5. History of smoking (≥ 10 pack years) -

Exclusion Criteria:

Volunteers will be excluded from the study if they meet any of the following criteria:

1. Uses oxygen continuously during daytime hours (nighttime use OK)
2. Requires > 10mg per day of prednisone (or equivalent corticosteroid dose) chronically
3. Concomitant presence of congestive heart failure, active coronary syndromes, or other disease that in the opinion of the investigator would increase the risk resulting from participation
4. Recent change in respiratory medications, including acute antibiotic or systemic corticosteroid interventions within the last 4 weeks
5. History of intolerance or hypersensitivity to hypertonic saline or short acting inhaled beta agonist
6. Significant broncho reactivity by examination or pulmonary function testing (PFT), that in the opinion of the investigator would increase the risk of HS use
7. Radiation exposure within the 12 months prior to study participation that would cause them to exceed Federal Regulations by participating in this study
8. Subjects with a positive pregnancy test
9. Subjects who, in the opinion of the Principal Investigator, should not participate in the study

Subjects may be temporarily excluded from screening should they experience a respiratory tract infection that requires treatment with antibiotics and/or steroids. They may become eligible for screening four weeks after completing their treatment providing their symptoms have resolved.

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Measure and compare the sustained effects on mucus clearance of two weeks of daily dosing of hypertonic saline versus a low salt control treatment for subjects with CB. | Approximately 11 weeks
  Using a gamma camera and inhalation of technicium bound to sulfur colloid, mucus clearance can be measured. Will do this with two different types of inhaled saline.

SECONDARY OUTCOMES:
We will also be collecting sputum and breath condensation to analyze for protein and inflammatory changes that might occur with exacerbations. | Within 2 years after all data collection has ended

OTHER OUTCOMES:
Changes in lung function testing (spirometry) | within 11 weeks of enrollment of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Ashley G Henderson, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No